CLINICAL TRIAL: NCT04888052
Title: Strength Muscular Assessment and Prolonged Preoperative Rehabilitation Interest in the Anterior Cruciate Ligament Rupture - a Preliminary Study
Brief Title: Prolonged Preoperative Rehabilitation in ACL Rupture.
Acronym: ISO-LCA-PREOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020_71; 2021-A00598-33 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-04-14; First posted 2021-05-17 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: Rehabilitation; preoperative; strength; isokinetic; anterior cruciate ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental)
  Interventions: Device: Acute ACL injury

INTERVENTIONS:
Device: Acute ACL injury — Quantification of the preoperative deficits, by an isokinetic dynamometer, in order to adapt the care management of patients found with a muscle deficiency. Patients with preoperative knee extensor deficits > 15% will benefit from an additional preoperative rehabilitation protocol (8 weeks).

SUMMARY:
Rupture of the anterior cruciate ligament is a serious and common injury. In young athletes, surgical reconstruction of the anterior cruciate ligament by autograft with hamstrings or patellar ligament is widely used.

Despite relatively standardized medical, surgical, and paramedical management, the results after ACL ligamentoplasty are not entirely satisfactory in term of return to sport. Recovery of the quadriceps strength is recognized as one of the decision-making criteria allowing the return to sport; however, significant muscle deficits are frequent at the time of return to sport.

If the postoperative management is well codified, focused on muscle strengthening and neuromuscular retraining, some studies have addressed the value of preoperative rehabilitation, and recommend a good preoperative muscular recovery of knee extensors and flexors, to obtain better postoperative results at the stage of the return to sports.

These results suggest that preoperative quadriceps strength should be considered as a predictor of the athletes' ability to return to sport activities.

It is estimated that around 10 to 30% of patients with preoperative deficits and could benefit from additional rehabilitation.

It can then be assumed that if the preoperative deficit is smaller, the postoperative deficit will also be smaller. This is the challenge of preoperative rehabilitation.

There are a few studies on preoperative rehabilitation which allow a gain in strength of knee extensors and flexors. However, the rehabilitation protocols applied to patients highly varied and there is no consensus on one protocol. The potential improvement is in the range of 10 to 20%.

The hypothesis of the study is that an optimal recovery of the strength of the preoperative knee extensors and flexors would reduce the postoperative deficit, thus improving the return to sport.

In the absence of reliable information on the frequency of muscle weakness in preoperative patients, we will conduct a preliminary study to obtain these data as well as the potential gain in strength with our preoperative rehabilitation protocol.

ELIGIBILITY:
Inclusion Criteria:

* Acute ACL injury (< 4 weeks) before surgical treatment
* Patient given written consent to participate in the study,
* Patient able to understand the protocol and willing to comply with its rules.
* Social security affiliated

Exclusion Criteria:

* Age < 18 years ou > 45 years,
* ACL rupture associated with fracture or complex meniscal tear or lesion to the lateral collateral ligament or posterior cruciate ligament
* History of ligament surgery on the affected and non-affected knee.
* fracture
* Isokinetic contraindications : cardiorespiratory, metabolic, neurological, cancer or hematological pathology contraindicating physical activity, long term steroid use (> 3 months), pregnancy, skin problems under load cell, osteoporosis, anticoagulants
* Patient under the protection of adults
* Informed consent not obtained

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 4-6 weeks after ACL injury
  Muscle strength: measurement of knee extensors and flexors peak torque on isokinetic dynamometer.

SECONDARY OUTCOMES:
Muscle strength | through study completion, an average of 20 weeks
  Muscle strength: measurement of knee extensors and flexors peak torque on isokinetic dynamometer.
Functional testing : SEBT | 4-6 weeks after ACL injury and through study completion, an average of 20 weeks
Title Questionnaires : Lyshom | 4-6 weeks after ACL injury and through study completion, an average of 20 weeks
Title Questionnaires : confidence questionnaire | 4-6 weeks after ACL injury and through study completion, an average of 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: André Thevenon, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Swynghedauw, Lille, France